CLINICAL TRIAL: NCT01637909
Title: Korean Life-Style Modification Effects on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0305
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Prehypertension; Hypertension
Keywords: Prehypertension, Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- general management (Active Comparator)
  Interventions: Drug: Control group who are advised for proper life style modification by the physician such as regular exercise and healthy diet without active intervention.
- The treatment group1 (Experimental): Korean DASH diet with sodium reduction intervention
  Interventions: Dietary Supplement: Treatment group 1(Dietary intervention)
- The treatment group2 (Experimental): Korean DASH diet with sodium reduction intervention and excersize intervention
  Interventions: Other: Treatment group 2(dietary and exercise intervention)

INTERVENTIONS:
Drug: Control group who are advised for proper life style modification by the physician such as regular exercise and healthy diet without active intervention. — All the study subjects will undergo baseline brachial blood pressure measurement(OMRON HEM 7080IT), central aortic blood pressure measurement with Sphygmocor device(AtCor Medical), baseline laboratory, 24hr urine Na measurement, 24 hour ambulatory blood pressure and cardiopulmonary exercise test. These tests will be repeated at the 8th week.
  Arms: general management
Dietary Supplement: Treatment group 1(Dietary intervention) — The dietary intervention is based on active education of the enrolled subjects based on Korean modified DASH diet. The enrolled subjects are advised to substitute processed white rice with whole grains such as barley. For protein, the subjects are advised to consume chicken and fish instead of red meat. Also, consumption of nuts are recommended where as processed foods containing high fructose corn syrup are not recommended. We will recommend to reduce salt intake by advising the subjects from adding table salts to their meals as well as adding salt during cooking. We will advise the subjects from eating pickles and condiments, which are the main source of salt in the Korean population. The degree of salt reduction before and after intervention will be assessed by 24 hour recall as well as measurement of 24 hour urine Na collection at baseline and at the 8th week. The compliance of the subjects will be assessed by 24hr recall as well.
  Arms: The treatment group1
Other: Treatment group 2(dietary and exercise intervention) — The dietary intervention will be combined with exercise intervention. At baseline, the subjects will undergo evaluation for (1) cardiopulmonary function by undergoing cardiopulmonary exercise test and 3 minute step test 2) muscle strength assessment by hand grip test and 3) push ups to assess muscle endurance. After the initial evaluation, the subjects will be subjected to a course in aerobic exercise and muscle strengthening exercise developed by the Yonsei University Physical education department and will receive an educational DVD program. The subjects will each be given an electronic step counter to assess the degree of exercise. All the subjects in the treatment group 2 will be advised to undergo moderate to stenuous aerobic exercise for least 150 minutes /per week. Also, the subjects will be educated to perform muscle strengthening exercise as specificed in the educational program. The subjects will be asked to submit an exercise diary to assess the degree of compliance.
  Arms: The treatment group2

SUMMARY:
In hypertension, lifestyle modification has been proven to be effective in reducing blood pressure while decreasing the risk of cardiovascular disease. The dietary approaches to stop hypertension(DASH) diet, sodium restriction and exercise has been shown to reduce systolic blood pressure by 8-14mmHg, 2-8mmHg and 4-9mmHg, respectively. The DASH-sodium diet has been shown to have additional systolic blood pressure lowering effect of 7.2mmHg, which is equal to adding one antihypertensive drug. However, as the dietary pattern is different in the Korean population, the investigators cannot implement the data from Western countries directly to the Korean population. For example, the consumption of dairy products is much smaller in the Korean population when compared to the western population. Therefore, the effectiveness of DASH-sodium diet and exercise on blood pressure lowering in the Korean population is not well defined. In this study, the investigators sought to determine the effectiveness of the DASH-salt diet and DASH-salt diet plus exercise on brachial blood pressure lowering. The study will be performed on untreated prehypertension patients and uncontrolled hypertensive patients undergoing anti hypertensive treatment with blood pressure measured between 140-159mmHg/90-99mmHg at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age >20
2. If the subject not taken antihypertension, SBP and DBP must be the following result.

   SBP: 120~159 mmHg , DBP: 80-99 mmHg
3. If the subject taken antihypertension, SBP and DBP must be the following result.

   SBP: 140-159mmHg ,DBP: 90-99 mmHg
4. BMI 18.5kg/m²~44kg/m²
5. Patients voluntarily agreed to participate in this study
6. Non-pregnant women, Non-breastfeeding women, women of childbearing age must be negative in HCG result.

(not taking an oral contraceptive)

Exclusion Criteria:

1. If the subject not taken antihypertension, SBP and DBP must be the following result.

   * 120>SBP>159 mmHg, 80>DBP>99 mmHg
2. If the subject taken antihypertension, the number of three or more antihypertensive
3. If the subject taken antihypertension, SBP and DBP must be the following result.

   * 140>SBP>159 mmHg, 90>DBP>99 mmHg
4. having the target organ disease, the following disease.

   * Heart disease: Lt.venricular hyperplasia, Angina, MI, Coronary revascularization, Heart failure
   * Brain disease: Stroke, TIA, Dementia
   * Kidney disease:
   * Pheripheral artery disease
   * Retinopathy Disease
5. Cancer, Liver disease
6. Regular drinking alcohol above 14 cup of during 1 week.
7. Pregnant women, Women of childbearing age tested positive in HCG result.
8. Pregnant women, Breastfeeding women
9. screening test result CS
10. illiteracy, a foreigner, the person who can't read the consent
11. the person who had participated other study in 3 months.
12. the person who inappropriate to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
changes of blood pressure after intervention | after 1 week, 4weeks, 8weeks intervention for each group intervention
  The primary outcome will be the difference in sitting brachial systolic blood pressure after 8 weeks intervention. The study population was determined by treatment group 1 will have systolic BP lowering effect of 11.5mmHg with standard deviation of 10.0mmHg and group 2 will have systolic BP lowering effect of 18.0mmHg with standard deviation of 15.0mmHg. with statistical power of 80% and drop out rate of 25%, the number needed was determined to be 32 in the control group, 22 in group 1 and 22 in group 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei universty medical center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee CJ, Kim JY, Shim E, Hong SH, Lee M, Jeon JY, Park S. The Effects of Diet Alone or in Combination with Exercise in Patients with Prehypertension and Hypertension: a Randomized Controlled Trial. Korean Circ J. 2018 Jul;48(7):637-651. doi: 10.4070/kcj.2017.0349. PMID 29968437